CLINICAL TRIAL: NCT03498768
Title: Epidemiology and Psychosocial Evaluation of Inpatient With Lung Opacity ：a Prospective Multicentre Study
Brief Title: Epidemiology and Psychosocial Evaluation of Inpatient With Lung Opacity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Principal Investigator, Clinical Professor, Peking University People's Hospital
Other Study IDs: PKUPH-DTS
Record Dates: First submitted 2018-04-05; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Psychological Distress
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatients with lung nodules: All inpatients in our department are invited to finish the questionnaire at inpatient education on the first day of hospitalization as the baseline date, then they are followed up by phone call to reevaluate their psychosocial status at 6 months and 1 year after the surgery.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Subjects will be invited to complete a detailed questionnaire regarding personal information, known risk factors for lung cancer and psychological status.

SUMMARY:
Lung cancer is one of the leading cause of cancer related death in China.Different from patients in the US, Chinese patients with lung nodules tend to be less related to smoking, and seem to be more willing to get operation despite of the doctors' suggestion of imaging surveillance.

This study is designed to figure out the risk factors for Chinese lung cancer patients and evaluate the psychosocial status of inpatients with lung nodules.

DETAILED DESCRIPTION:
Smoking is the only determinate risk factor proposed by the NCCN（National Comprehensive Cancer Network） Clinical Practice Guidelines for lung cancer screening. However, it has been estimated that over half of Chinese female lung cancer patients are non-smokers. Thus it might be reasonable to take unique Chinese cooking habit and environment pollution into consideration when it comes to the risk factors for lung cancer in Chinese people.

Lung nodules are reported to exist in 25-70% patients who have undergone LDCT （Low-dose Computed Tomography）examination. However, the prevalence of malignant nodules is reported to be 1.1-3% by different researchers. Even in country with comprehensive medical consulting system and lung nodule management consensus, almost all patients assume their lung nodules to be malignant when detected by LDCT for the first time.The investigators noticed nearly 1/3 of the inpatients are determined to get operation despite the surgeons' suggestion of CT surveillance according to the NCCN guideline in Department of Thoracic surgery in Peking University People's Hospital. As there's no evidence suggesting lung nodules in Chinese people have more possibility of malignancy, the investigators would like to know whether those patients who choose to get operation "ahead of the guideline" has higher level of cancer distress, and figure out whether psychosocial factors should be taken into consideration of lung nodules management when living with an indeterminate tumor has added up to patients' negative emotion and reduced their quality of life.

The investigators do the survey on the first day of admission during the inpatient education, help patients fill in the questionnaire including personal information, smoking history, medical history, their diet and lifestyle habits, family history of malignant neoplasm, any past or current environmental exposures and psychological status.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in Department of Thoracic Surgery in Peking University People's Hospital and Beijing Haidian Hospital.
* Tolerant to surgery with accessible pathology outcome.
* Aged between 18-80.
* Signed Informed Consent Form.

Exclusion Criteria:

* Patients who have difficulty in reading and writing.
* Poor physical status without sufficient respiratory reserve to undergo surgery.
* Unaccessible for surveillance after surgery.
* Refuse to take part.
* Other circumstances which is deemed inappropriate for enrollment by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients aged between 18-80, tolerant to surgery with accessible pathology outcome are eligible.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Risk factors for Chinese lung cancer patients | 1.5 years
  Patients with lung nodules are invited to fill in a questionnaire including personal information, smoking history, medical history, their diet and lifestyle habits, family history of malignant neoplasm, this procedure is finished during inpatient education before the operation. After the operation, we analyze the factors and patients' pathology results to figure out the risk factors for Chinese lung cancer patients.
Psychological status of patients with lung nodules | 1.5 years
  Patients with lung nodules are invited to fill in the Hospital Anxiety and Depression Scale (HADS) during inpatient education. Patients are thus grouped depending on whether they have indication for biopsy or operation according to the NCCN guideline for lung nodules management. As a result, patients who accept surveillance long enough or have proper indication for operation are one group, patients who stop surveillance and choose to get operation "ahead of time" are the other group. The level of negative emotion would be analyzed and compared afterwards.

SECONDARY OUTCOMES:
Life quality of patients with lung nodules | 1.5 years
  Patients with lung nodules are invited to fill in the MOS item short from health survey (SF-36) scale during inpatient education. Patients are thus grouped depending on whether they have indication for biopsy or operation according to the NCCN guideline for lung nodules management. As a result, patients who accept surveillance long enough or have proper indication for operation are one group, patients who stop surveillance and choose to get operation "ahead of time" are the other group. The quality of life would be analyzed and compared afterwards.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, MM, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China